CLINICAL TRIAL: NCT03740919
Title: A Prospective, Randomized, Double-Blind Comparison of LY900014 to Humalog With an Open-Label Postprandial LY900014 Treatment Group in Children and Adolescents With Type 1 Diabetes
Brief Title: A Study Comparing LY900014 to Insulin Lispro (Humalog) in Children and Adolescents With Type 1 Diabetes
Acronym: PRONTO-Peds
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16698; I8B-MC-ITSB (Other: Eli Lilly and Company); 2018-002371-18 (EudraCT Number)
Record Dates: First submitted 2018-11-12; First posted 2018-11-14 (Actual); Results first posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2021-12

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: prandial insulin; multiple daily injections; pediatric patients; postmeal dosing
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro; Insulin Glargine; insulin degludec

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Insulin Lispro (Humalog) (Active Comparator): Participants received 100 units per milliliter (U/mL) insulin lispro (Humalog) administered subcutaneously (SC), 0 to 2 minutes before each meal with once or twice daily basal insulin. Preprandial insulin doses were individualized and titrated according to protocol-defined targets.
  Interventions: Drug: Insulin Lispro; Drug: Insulin Glargine; Drug: Insulin Degludec
- LY900014 (Experimental): Participants received 100 U/mL LY900014 administered SC, 0 to 2 minutes before start of the meal.
  Interventions: Drug: LY900014
- LY900014 Postmeal (Experimental): Participants received 100 U/mL LY900014 administered SC, up to 20 minutes after the start of the meal.
  Interventions: Drug: LY900014

INTERVENTIONS:
Drug: LY900014 — Administered SC
  Other Names: Ultra-Rapid Lispro
  Arms: LY900014; LY900014 Postmeal
Drug: Insulin Lispro — Administered SC
  Other Names: Humalog; LY275585
  Arms: Insulin Lispro (Humalog)
Drug: Insulin Glargine — Administered SC
  Arms: Insulin Lispro (Humalog)
Drug: Insulin Degludec — Administered SC
  Arms: Insulin Lispro (Humalog)

SUMMARY:
The reason for this study is to compare the study drug LY900014 to insulin lispro (Humalog) in children and adolescents with type 1 diabetes (T1D).

ELIGIBILITY:
Inclusion Criteria:

* T1D for at least 6 months at the screening visit.
* Have been treated with only one of the following rapid-acting insulin analogs as part of an multiple daily injection regimen for at least the last 90 days prior to the screening visit:

  * insulin lispro U-100, or
  * insulin aspart
  * insulin glulisine or
  * fast acting insulin aspart
* Have been treated with only one of the following basal insulins for at least the last 90 days prior to the screening visit:

  * insulin glargine U-100 (once a day [QD] or twice a day [BID]), or
  * insulin detemir U-100 (QD or BID), or
  * insulin degludec U-100 (QD)
* Have a HbA1c value ≤ 9.9% at the screening visit.

Exclusion Criteria:

* Have current hypoglycemic unawareness or have had more than 1 episode of severe hypoglycemia within 6 months prior to the screening visit.
* Have had more than 1 emergency room visit or hospitalization due to poor glucose control within 6 months prior to the screening visit.
* Have been on a treatment regimen that includes regular human insulin, neutral protamine Hagedorn (NPH), Afrezza® (insulin human) inhalation powder, any premixed insulins or use of diluted insulins within 90 days prior to the screening visit.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 751 (Actual)
Dates: Start 2019-04-07 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (111):
- United States (27):
  - University of Alabama Birmingham, Birmingham, Alabama
  - University of Arizona, Tucson, Arizona
  - Children's Hospital Los Angeles - Dept of Endocrinology, Los Angeles, California
  - Stanford University School of Medicine - Division of Pediatric Endocrinology & Diabetes, Palo Alto, California
  - Center of Excellence in Diabetes & Endocrinology, Sacramento, California
  - Rady Childrens Hospital - San Diego, San Diego, California
  - Barbara Davis Center, Aurora, Colorado
  - Florida Hospital, Orlando, Florida
  - Tallahassee Memorial HealthCare, Tallahassee, Florida
  - University of South Florida Diabetes & Endocrinology Center, Tampa, Florida
  - VanMeter Pediatric Endocrinology, P.C., Atlanta, Georgia
  - St. Luke's Children's Endocrinology, Boise, Idaho
  - Rocky Mountain Diabetes and Osteoporosis Center, Idaho Falls, Idaho
  - Indiana University- Riley Children's Hospital, Indianapolis, Indiana
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Barry Reiner Clinic, Baltimore, Maryland
  - Joslin Diabetes Center, Boston, Massachusetts
  - Children's Mercy Hospital, Kansas City, Missouri
  - UBMD Pediatrics, Buffalo, New York
  - Suny Health Science Center at Syracuse, Syracuse, New York
  - Endocrinology Services NorthWest, Bend, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Diabetes & Endocrinology, P.A., Austin, Texas
  - Texas Institute for Kidney and Endocrine Disorders, Lufkin, Texas
  - Diabetes and Glandular Disease Research Associates PA, San Antonio, Texas
  - MultiCare Institute for Research & Innovation, Tacoma, Washington
- Austria (2):
  - Universitätsklinikum Graz, Graz, Styria
  - Universitätsklinik Innsbruck, Innsbruck, Tyrol
- Brazil (3):
  - Hospital das Clinicas da FMRP, Ribeirão Preto, São Paulo
  - CPCLIN, São Paulo, São Paulo
  - CPQuali Pesquisa Clínica, São Paulo
- China (6):
  - Children's hospital of Nanjing, Nanjing, Jiangsu
  - Wuxi Children's Hospital, Wuxi, Jiangsu
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin, Nangang District
  - Children's Hospital Capital Institute of Pediatrics, Beijing
  - Children's hospital of Fudan University, Shanghai
  - Zhengzhou Children's Hospital, Zhengzhou
- Czechia (6):
  - Fakultni Nemocnice v Motole, Prague, Motole
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Pediatricke odd. Nemocnice Jihlava, Jihlava
  - Medica Iberia, Opava
  - FN Ostrava, Ostrava-Poruba
  - Pardubicka krajska nemocnice, Pardubice
- Herlev and Gentofte Hospital, Herlev, Denmark
- France (4):
  - CHRU Lille - Hôpital Jeanne de Flandre, Lille
  - CHU Hopital d'enfants de la Timone, Marseille
  - Hopital Robert Debre, Paris
  - Hôpital Universitaire Necker enfants malades, Paris
- Germany (4):
  - InnoDiab Forschung Gmbh, Essen, North Rhine-Westphalia
  - Diabetologische Schwerpunktpraxis Dr. Ziegler, Münster, North Rhine-Westphalia
  - Medizinisches Versorgungszentrum am Universitätsklinikum Leipzig GmbH, Leipzig, Saxony
  - RED-Institut GmbH, Oldenburg in Holstein, Schleswig-Holstein
- Israel (5):
  - Shamir Medical Center (Asaf Harofe)-Pediatric Endocrinology Unit, Beer Yaakov
  - Soroka Medical Center - Pediatric Outpatient Clinic, Beersheba
  - Rambam Medical Center - Department of Pediatrics A, Ruth Rappaport Children's Hospital, Haifa
  - Schneider Children's Medical Center, Petah Tikva
  - Shiba Medical Center, Ramat Gan
- Italy (6):
  - Azienda Ospedaliera Umberto I, Ancona
  - Azienda Ospedaliero Universitaria Meyer, Florence
  - IRCCS Ospedale San Raffaele, Milan
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Ospedale Bambino Gesu, Roma
  - Ospedale Civile Maggiore Borgo Trento, Verona
- Japan (6):
  - Saitama Children's Medical Center, Saitama-shi, Saitama
  - Nihon University Hospital, Chiyoda-ku, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku-ku, Tokyo
  - Hiroshima Prefectural Hospital, Hiroshima
  - Niigata University Medical & Dental Hospital, Niigata
  - Osaka City University Hospital, Osaka
- Mexico (5):
  - Unidad de Investigacion Clinica Cardiometabolica de Occidente, Guadalajara, Jalisco
  - Centro de Inv. Medica de Occidente, SC, Zapopan, Jalisco
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey, N.L.
  - Cli-nica Hospital Cemain, Tampico, Tamaulipas
  - Hospital Angeles Puebla, Puebla City
- Poland (3):
  - Gdanski Uniwersytet Medyczny, Gdansk
  - Uniwersytecki Szpital Kliniczny, Lodz
  - Instytut Diabetologii Sp. z o.o, Warsaw
- Puerto Rico (2):
  - Pediatric Endocrine Research Associates, Rio Piedras, PR
  - San Jorge Children and Women's Hospital- Shipping Location, San Juan, PR
- Russia (9):
  - Research Institute for Pediatric Endocrinology, Moscow
  - Morozovsky Children's City Clinical Hospital, Moscow
  - St.Petersburg Children's City Polyclinic #44, Saint Petersburg
  - Samarskiy Regional Children's Clinical Hospital, Samara
  - Saratov State Medical University, Saratov
  - Smolensk Regional Children's Clinical Hospital, Smolensk
  - Siberian State Medical University of Roszdrav, Tomsk
  - Tver Children's Clinical Hospital, Tver'
  - Voronezh State Medical University, Voronezh
- Spain (9):
  - Hospital Virgen del Camino, Pamplona, Navarre
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - CHUS - Hospital Clinico Universitario, A Coruña
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario HM Monteprincipe, Boadilla del Monte
  - Hospital Sant Joan de Déu, Esplugues de Llobregat
  - Clínica nuevas Tecnologías en Diabetes y Endocrinología (NTDE), Seville
  - Hospital Universitario La Fe de Valencia, Valencia
  - Hospital Txagorritxu, Vitoria-Gasteiz
- Ukraine (6):
  - Ivano-Frankivsk regional clinical children hospital, Ivano-Frankivsk
  - Institute of the Health Care of Children & Adolescents, Kharkiv
  - V.P. Komisarenko Institute of Endocrinology and Metabolism of NAMS of Ukraine, Kyiv
  - Odesa regional children's clinical hospital, Odesa
  - Vinnytsia Regional Clinical Highly Specialized Endocrinology Center, Vinnytsia
  - Zaporizhzhia regional clinical children hospital, Zaporizhzhia
- United Kingdom (7):
  - Stepping Hill Hospital, Stockport, Cheshire
  - Norfolk and Norwich Hospital, Norwich, Norfolk
  - King's Mill Hospital, Sutton in Ashfield, Nottinghamshire
  - Worthing Hospital, Worthing, West Sessex
  - St Richards Hospital, Chichester, West Sussex
  - St James's University Hospital, Leeds, West Yorkshire
  - St. George's University Hospitals NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: A Study Comparing LY900014 to Insulin Lispro (Humalog) in Children and Adolescents With Type 1 Diabetes — https://trials.lillytrialguide.com/en-US/trial/3msKrLw2I0WuYqosKQw22Q

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study included a 4-week lead-in period using open-label insulin lispro (Humalog) followed by a 26-week double-blind treatment period (LY900014 and Insulin Lispro) and one Open-label treatment arm (LY900014 Postmeal).
Pre-assignment Details: The purpose of the lead-in period was to obtain blood glucose (BG) values along with basal and prandial insulin doses to assess basal and mealtime insulin dosing and to determine baseline hypoglycemia rates.
Groups:
- Insulin Lispro (Humalog) Lead-in: Participants were switched to open-label insulin lispro (Humalog) administered subcutaneously (SC), using a unit for unit conversion or the dose could have been determined based on investigator's clinical judgement.
- Insulin Lispro (Humalog): Participants received 100 units per milliliter (U/mL) insulin lispro (Humalog) administered SC, 0 to 2 minutes before each meal with once or twice daily basal insulin. Preprandial insulin doses were individualized and titrated according to protocol-defined targets.
- LY900014: Participants received 100 U/mL LY900014 administered SC 0 to 2 minutes before start of the meal.
- LY900014 Postmeal: Participants received 100 U/mL LY900014 administered SC up to 20 minutes after the start of the meal.
Period: Lead-in Period
Arm/Group | Insulin Lispro (Humalog) Lead-in | Insulin Lispro (Humalog) | LY900014 | LY900014 Postmeal
Started | 751 | 0 | 0 | 0
Received at Least One Dose of Study Drug | 751 | 0 | 0 | 0
Completed | 716 | 0 | 0 | 0
Not Completed | 35 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 10 | 0 | 0 | 0
Not completed — Due to Coronavirus Disease 2019 (COVID-19) | 18 | 0 | 0 | 0
Not completed — Study Task Too Burdensome | 1 | 0 | 0 | 0
Not completed — Lab Results Did Not Match Inclusion Criteria | 1 | 0 | 0 | 0
Not completed — Withdrew Consent Due to Required Procedures | 1 | 0 | 0 | 0
Period: Treatment Period
Arm/Group | Insulin Lispro (Humalog) Lead-in | Insulin Lispro (Humalog) | LY900014 | LY900014 Postmeal
Started (After completion of Lead-in Period, participants were randomized to either blinded LY900014 or Humalog or open-label LY900014.) | 0 | 298 (Participants were randomized from Lead-in Period to Insulin Lispro (Humalog).) | 280 (Participants were randomized from Lead-in Period to LY900014.) | 138 (Participants were randomized from Lead-in Period to open-label LY900014.)
Received at Least One Dose of Study Drug | 0 | 298 | 280 | 138
Completed | 0 | 288 | 266 | 135
Not Completed | 0 | 10 | 14 | 3
Not completed — Adverse Event | 0 | 0 | 2 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 7 | 6 | 2
Not completed — Terminated by Sponsor | 0 | 1 | 0 | 0
Not completed — Issue with Insulin Pump | 0 | 1 | 0 | 0
Not completed — Due to COVID-19 Pandemic | 0 | 0 | 3 | 1
Not completed — Failure of Inclusion Criteria | 0 | 0 | 1 | 0
Not completed — Not Completing Diary | 0 | 0 | 1 | 0
Not completed — Insulin Painful to Participant | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who were randomly assigned to study treatment..
Groups:
- Insulin Lispro (Humalog): Participants received 100 U/mL insulin lispro (Humalog) administered SC, 0 to 2 minutes before each meal with once or twice daily basal insulin. Preprandial insulin doses were individualized and titrated according to protocol-defined targets.
- Total: Total of all reporting groups
Arm/Group | Insulin Lispro (Humalog) | LY900014 | LY900014 Postmeal | Total
Number analyzed (Participants) | 298 | 280 | 138 | 716
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.4 (3.2) | 12.1 (3.4) | 12.3 (3.8) | 12.3 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140 | 144 | 65 | 349
  Male | 158 | 136 | 73 | 367
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 6 | 0 | 12
  Asian | 20 | 13 | 7 | 40
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 2
  Black or African American | 7 | 3 | 1 | 11
  White | 256 | 256 | 126 | 638
  More than one race | 4 | 0 | 1 | 5
  Unknown or Not Reported | 3 | 2 | 3 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 51 | 55 | 25 | 131
  Czechia | 26 | 23 | 11 | 60
  Japan | 7 | 3 | 2 | 12
  Ukraine | 57 | 53 | 27 | 137
  United Kingdom | 3 | 5 | 2 | 10
  Spain | 21 | 19 | 8 | 48
  Russia | 23 | 21 | 12 | 56
  Austria | 1 | 0 | 0 | 1
  China | 11 | 7 | 4 | 22
  Brazil | 22 | 20 | 13 | 55
  Poland | 14 | 13 | 6 | 33
  Denmark | 0 | 1 | 0 | 1
  Italy | 15 | 15 | 6 | 36
  Mexico | 25 | 22 | 11 | 58
  Israel | 15 | 15 | 5 | 35
  France | 1 | 1 | 2 | 4
  Germany | 6 | 7 | 4 | 17
HbA1c at Baseline [Mean (Standard Deviation); unit: percentage of HbA1c] | 7.81 (0.91) | 7.81 (0.87) | 7.77 (0.85) | 7.80 (0.88)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) Efficacy Estimand at Week 26
Description: Change from baseline in HbA1c was analyzed using mixed model repeated measures (MMRM) and includes fixed class effects of treatment, strata (pooled country, type of basal insulin, and age group), visit, and treatment-by-visit interaction, as well as the continuous, fixed covariates of baseline value. An unstructured covariance structure will be used to model the within-participant errors.
  The Efficacy estimand included data collected prior to permanent discontinuation of study drug through Week 26.
Time Frame: Baseline, Week 26
Population: All participants randomly assigned to study drug with baseline and at least one postbaseline measurement available while on study drug, per protocol.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Insulin Lispro (Humalog) | LY900014
Number analyzed (Participants) | 280 | 260
percentage of HbA1c | 0.09 (0.052) | 0.06 (0.054)
Statistical Analysis 1: Comparison: Insulin Lispro (Humalog) vs LY900014; Test type: Non-Inferiority — Noninferiority margin [NIM]=0.4% for HbA1c; p = 0.783, Mixed Models Analysis; Least Squares (LS) Mean Difference = -0.02, 95% CI 2-sided [-0.17 to 0.13]

2. Secondary Outcome: Change From Baseline in HbA1c (Postprandial) at Week 26
Description: Change from baseline in HbA1c postprandial was analyzed using (MMRM and includes fixed class effects of treatment, strata (pooled country, type of basal insulin, and age group), visit, and treatment-by-visit interaction, as well as the continuous, fixed covariates of baseline value. An unstructured covariance structure will be used to model the within-participant errors.
  The Efficacy estimand included data collected prior to permanent discontinuation of study drug through Week 26.
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Insulin Lispro (Humalog) | LY900014 Postmeal
Number analyzed (Participants) | 280 | 131
percentage of HbA1c | 0.09 (0.052) | 0.07 (0.076)
Statistical Analysis 1: Comparison: Insulin Lispro (Humalog) vs LY900014 Postmeal; Test type: Non-Inferiority — NIM of 0.4%; p = 0.867, Mixed Models Analysis; LS Mean Difference = -0.02, 95% CI 2-sided [-0.20 to 0.17]

3. Secondary Outcome: Percentage of Participants With Documented Post-dose Hypoglycemic Events Within 1 and 2 Hours After the Prandial Dose
Description: Documented post-dose hypoglycemia <54 milligrams per deciliter (mg/dL) and ≤ 70 mg/dL that occurred 1 and 2 hours after prandial dose.
Time Frame: Baseline through Week 26
Population: All randomized participants who received at least one dose of the randomly assigned study drug with non-missing baseline value and at least one non-missing post-baseline value of the response variable.
Measure: Least Squares Mean (Standard Error); unit: percentage of participants
Arm/Group | Insulin Lispro (Humalog) | LY900014 | LY900014 Postmeal
Number analyzed (Participants) | 298 | 280 | 138
percentage of participants
  <54 mg/dL 1 Hour Post Dose | 26.50 (2.563) | 36.79 (2.891) | 29.70 (3.897)
  <54 mg/dL 2 Hour Post Dose | 54.04 (2.896) | 63.61 (2.883) | 57.88 (4.216)
  ≤70 mg/dL 1 Hour Post Dose | 49.67 (2.901) | 63.92 (2.874) | 48.51 (4.261)
  ≤70 mg/dL 2 Hour Post Dose | 77.03 (2.449) | 82.67 (2.267) | 70.29 (3.912)
Statistical Analysis 1: Comparison: Insulin Lispro (Humalog) vs LY900014; < 54 mg/dL 1 hour post-dose; Test type: Superiority; p = 0.008, Regression, Logistic; Odds Ratio (OR) = 1.61, 95% CI 2-sided [1.13 to 2.30]
Statistical Analysis 2: Comparison: Insulin Lispro (Humalog) vs LY900014 Postmeal; < 54 mg/dL 1 hour post-dose; Test type: Superiority; p = 0.487, Regression, Logistic; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.75 to 1.83]
Statistical Analysis 3: Comparison: LY900014 vs LY900014 Postmeal; < 54 mg/dL 1 hour post-dose; Test type: Superiority; p = 0.153, Regression, Logistic; Odds Ratio (OR) = 0.73, 95% CI 2-sided [0.47 to 1.13]
Statistical Analysis 4: Comparison: Insulin Lispro (Humalog) vs LY900014; < 54 mg/dL 2 hour post-dose; Test type: Superiority; p = 0.020, Regression, Logistic; Odds Ratio (OR) = 1.49, 95% CI 2-sided [1.06 to 2.08]
Statistical Analysis 5: Comparison: Insulin Lispro (Humalog) vs LY900014 Postmeal; < 54 mg/dL 2 hour post-dose; Test type: Superiority; p = 0.455, Regression, Logistic; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.78 to 1.76]
Statistical Analysis 6: Comparison: LY900014 vs LY900014 Postmeal; < 54 mg/dL 2 hour post-dose; Test type: Superiority; p = 0.259, Regression, Logistic; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.52 to 1.19]
Statistical Analysis 7: Comparison: Insulin Lispro (Humalog) vs LY900014; ≤ 70 mg/dL 1 hour post-dose; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.79, 95% CI 2-sided [1.29 to 2.51]
Statistical Analysis 8: Comparison: Insulin Lispro (Humalog) vs LY900014 Postmeal; ≤ 70 mg/dL 1 hour post-dose; Test type: Superiority; p = 0.822, Regression, Logistic; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.64 to 1.43]
Statistical Analysis 9: Comparison: LY900014 vs LY900014 Postmeal; ≤ 70 mg/dL 1 hour post-dose; Test type: Superiority; p = 0.003, Regression, Logistic; Odds Ratio (OR) = 0.53, 95% CI 2-sided [0.35 to 0.80]
Statistical Analysis 10: Comparison: Insulin Lispro (Humalog) vs LY900014; ≤ 70 mg/dL 2 hour post-dose; Test type: Superiority; p = 0.092, Regression, Logistic; Odds Ratio (OR) = 1.42, 95% CI 2-sided [0.94 to 2.14]
Statistical Analysis 11: Comparison: Insulin Lispro (Humalog) vs LY900014 Postmeal; ≤ 70 mg/dL 2 hour post-dose; Test type: Superiority; p = 0.133, Regression, Logistic; Odds Ratio (OR) = 0.71, 95% CI 2-sided [0.45 to 1.11]
Statistical Analysis 12: Comparison: LY900014 vs LY900014 Postmeal; ≤ 70 mg/dL 2 hour post-dose; Test type: Superiority; p = 0.004, Regression, Logistic; Odds Ratio (OR) = 0.50, 95% CI 2-sided [0.31 to 0.80]

4. Secondary Outcome: Rate of Documented Post-dose Hypoglycemic Events Within 1 and 2 Hours After the Prandial Dose
Description: Documented post-dose hypoglycemia event is an event of blood glucose of < 54 mg/dL and ≤70 mg/dL that occurred within 1 and 2 hours after the prandial dose. The rate of documented hypoglycemia was estimated by a negative binomial regression including treatment and age group as independent variable and number of episodes as dependent variables with log (exposure/365.25 days) as the offset in the model.
Time Frame: Baseline through Week 26
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Events per participant per year
Arm/Group | Insulin Lispro (Humalog) | LY900014 | LY900014 Postmeal
Number analyzed (Participants) | 298 | 280 | 138
Events per participant per year
  < 54mg/dL 1 Hour Post Dose | 1.59 (0.251) | 2.04 (0.262) | 1.38 (0.287)
  < 54 mg/dL 2 Hour Post Dose | 4.48 (0.454) | 5.95 (0.510) | 6.17 (0.816)
  ≤70 mg/dL 1 Hour Post Dose | 6.54 (1.036) | 8.46 (0.992) | 5.29 (1.145)
  ≤70 mg/dL 2 Hour Post Dose | 19.0 (1.58) | 23.7 (1.86) | 21.1 (2.31)
Statistical Analysis 1: Comparison: Insulin Lispro (Humalog) vs LY900014; < 54 mg/dL 1 hour post-dose; Test type: Superiority; p = 0.220, Negative binomial regression; Treatment and age group as covariates, log (exposure/365.25 days) as the offset in the model
Statistical Analysis 2: Comparison: Insulin Lispro (Humalog) vs LY900014 Postmeal; < 54 mg/dL 1 hour post-dose; Test type: Superiority; p = 0.599, Negative binomial regression; Treatment and age group as covariates, log (exposure/365.25 days) as the offset in the model
Statistical Analysis 3: Comparison: LY900014 vs LY900014 Postmeal; < 54 mg/dL 1 hour post-dose; Test type: Superiority; p = 0.112, Negative binomial regression; Treatment and age group as covariates, log (exposure/365.25 days) as the offset in the model
Statistical Analysis 4: Comparison: Insulin Lispro (Humalog) vs LY900014; < 54 mg/dL 2 hour post-dose; Test type: Superiority; p = 0.034, Negative binomial regression; Treatment and age group as covariates, log (exposure/365.25 days) as the offset in the model
Statistical Analysis 5: Comparison: Insulin Lispro (Humalog) vs LY900014 Postmeal; < 54 mg/dL 2 hour post-dose; Test type: Superiority; p = 0.055, Negative binomial regression; Treatment and age group as covariates, log (exposure/365.25 days) as the offset in the model
Statistical Analysis 6: Comparison: LY900014 vs LY900014 Postmeal; < 54 mg/dL 2 hour post-dose; Test type: Superiority; p = 0.814, Negative binomial regression; Treatment and age group as covariates, log (exposure/365.25 days) as the offset in the model
Statistical Analysis 7: Comparison: Insulin Lispro (Humalog) vs LY900014; ≤70 mg/dL 1 hour post-dose; Test type: Superiority; p = 0.194, Negative binomial regression
Statistical Analysis 8: Comparison: Insulin Lispro (Humalog) vs LY900014 Postmeal; ≤70 mg/dL 1 hour post-dose; Test type: Superiority; p = 0.428, Negative binomial regression; Treatment and age group as covariates, log (exposure/365.25 days) as the offset in the model
Statistical Analysis 9: Comparison: LY900014 vs LY900014 Postmeal; ≤70 mg/dL 1 hour post-dose; Test type: Superiority; p = 0.057, Negative binomial regression; Treatment and age group as covariates, log (exposure/365.25 days) as the offset in the model
Statistical Analysis 10: Comparison: Insulin Lispro (Humalog) vs LY900014; ≤70 mg/dL 2 hour post-dose; Test type: Superiority; p = 0.056, Negative binomial regression; Treatment and age group as covariates, log (exposure/365.25 days) as the offset in the model
Statistical Analysis 11: Comparison: Insulin Lispro (Humalog) vs LY900014 Postmeal; ≤70 mg/dL 2 hour post-dose; Test type: Superiority; p = 0.435, Negative binomial regression; Treatment and age group as covariates, log (exposure/365.25 days) as the offset in the model
Statistical Analysis 12: Comparison: LY900014 vs LY900014 Postmeal; ≤70 mg/dL 2 hour post-dose; Test type: Superiority; p = 0.404, Negative binomial regression; Treatment and age group as covariates, log (exposure/365.25 days) as the offset in the model

5. Secondary Outcome: Percentage of Participants With Documented Hypoglycemic Events
Description: Documented hypoglycemia is defined as <54 mg/dL and ≤70 mg/dL, respectively.
Time Frame: Baseline through Week 26
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percentage of participants
Arm/Group | Insulin Lispro (Humalog) | LY900014 | LY900014 Postmeal
Number analyzed (Participants) | 298 | 280 | 138
percentage of participants
  <54 mg/dL | 80.81 (2.283) | 81.37 (2.329) | 74.45 (3.718)
  ≤70 mg/dL | 93.98 (1.375) | 92.55 (1.569) | 87.62 (2.806)
Statistical Analysis 1: Comparison: Insulin Lispro (Humalog) vs LY900014; <54 mg/dL; Test type: Superiority; p = 0.864, Regression, Logistic; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.68 to 1.57]
Statistical Analysis 2: Comparison: Insulin Lispro (Humalog) vs LY900014 Postmeal; <54 mg/dL; Test type: Superiority; p = 0.132, Regression, Logistic; Odds Ratio (OR) = 0.69, 95% CI 2-sided [0.43 to 1.12]
Statistical Analysis 3: Comparison: LY900014 vs LY900014 Postmeal; Test type: Superiority; p = 0.104, Regression, Logistic; Odds Ratio (OR) = 0.67, 95% CI 2-sided [0.41 to 1.09]
Statistical Analysis 4: Comparison: Insulin Lispro (Humalog) vs LY900014; ≤70 mg/dL; Test type: Superiority; p = 0.489, Regression, Logistic; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.42 to 1.52]
Statistical Analysis 5: Comparison: Insulin Lispro (Humalog) vs LY900014 Postmeal; ≤70 mg/dL; Test type: Superiority; p = 0.025, Regression, Logistic; Odds Ratio (OR) = 0.45, 95% CI 2-sided [0.23 to 0.90]
Statistical Analysis 6: Comparison: LY900014 vs LY900014 Postmeal; ≤70 mg/dL; Test type: Superiority; p = 0.099, Regression, Logistic; Odds Ratio (OR) = 0.57, 95% CI 2-sided [0.29 to 1.11]

6. Secondary Outcome: Rate of Documented Hypoglycemia Events
Description: Documented hypoglycemia is defined as a hypoglycemic event of blood glucose of ≤70 mg/dL or <54 mg/dL. The rate of documented hypoglycemia was estimated by negative binomial regression including treatment and age group as independent variables and number of episodes as dependent variable with log (exposure/365.25 days) as the offset in the model.
Time Frame: Week 0 through Week 26
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: events per participant per year
Arm/Group | Insulin Lispro (Humalog) | LY900014 | LY900014 Postmeal
Number analyzed (Participants) | 298 | 280 | 138
events per participant per year
  < 54 mg/dL | 16.6 (1.23) | 16.1 (1.20) | 17.7 (1.99)
  ≤70 mg/dL | 78.0 (4.23) | 75.1 (4.44) | 76.1 (6.10)
Statistical Analysis 1: Comparison: Insulin Lispro (Humalog) vs LY900014; < 54 mg/dL; Test type: Superiority; p = 0.732, Negative binomial regression
Statistical Analysis 2: Comparison: Insulin Lispro (Humalog) vs LY900014 Postmeal; < 54 mg/dL; Test type: Superiority; p = 0.638, Negative binomial regression
Statistical Analysis 3: Comparison: LY900014 vs LY900014 Postmeal; <54 mg/dL; Test type: Superiority; p = 0.462, Negative binomial regression
Statistical Analysis 4: Comparison: Insulin Lispro (Humalog) vs LY900014; ≤ 70 mg/dL; Test type: Superiority; p = 0.632, Negative binomial regression
Statistical Analysis 5: Comparison: Insulin Lispro (Humalog) vs LY900014 Postmeal; ≤ 70 mg/dL; Test type: Superiority; p = 0.800, Negative binomial regression
Statistical Analysis 6: Comparison: LY900014 vs LY900014 Postmeal; ≤ 70 mg/dL; Test type: Superiority; p = 0.889, Negative binomial regression

7. Secondary Outcome: Rate of Severe Hypoglycemia
Description: Severe hypoglycemia: during these episodes, participants have an altered mental status and cannot assist in their own care, may be semiconscious or unconscious, or experience coma with or without seizures, and require assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions.
  The rate of severe hypoglycemia per 100 years was calculated as: 100 times the total number of severe hypoglycemia episodes within the period divided by total exposure (in year) for all participants within the treatment group.
Time Frame: Week 0 through Week 26
Population: as for outcome 3
Measure: Number; unit: Events per participant per 100 years
Arm/Group | Insulin Lispro (Humalog) | LY900014 | LY900014 Postmeal
Number analyzed (Participants) | 298 | 280 | 138
Events per participant per 100 years | 2.05 | 2.20 | 0.00

8. Secondary Outcome: Change From Baseline in Insulin Dose at Week 26
Description: Change from baseline in insulin dose was analyzed using mixed model repeated measures (MMRM) and includes fixed class effects of treatment, strata (pooled country, type of basal insulin, age group, and HbA1c stratum (≤8.0%, >8.0%)), baseline value, visit and treatment-by-visit interaction. An unstructured covariance structure was used to model the within-participant errors.
Time Frame: Baseline, Week 26
Population: All participants randomly assigned to study drug with baseline and at least one postbaseline measurement available while on study drug.
Measure: Least Squares Mean (Standard Error); unit: Unit per day
Arm/Group | Insulin Lispro (Humalog) | LY900014 | LY900014 Postmeal
Number analyzed (Participants) | 283 | 264 | 132
Unit per day
  Total Daily Basal Insulin Dose | 2.3 (0.28) | 2.9 (0.29) | 2.7 (0.40)
  Total Daily Insulin Dose: number analyzed (Participants) | 279 | 256 | 131
  Total Daily Insulin Dose | 5.3 (0.66) | 5.8 (0.69) | 5.0 (0.96)
Statistical Analysis 1: Comparison: Insulin Lispro (Humalog) vs LY900014; Total Daily Basal Insulin; Test type: Superiority; p = 0.130, Mixed Models Analysis; LS Mean Difference = 0.6, 95% CI 2-sided [-0.2 to 1.4]
Statistical Analysis 2: Comparison: Insulin Lispro (Humalog) vs LY900014 Postmeal; Total Daily Basal Insulin; Test type: Superiority; p = 0.404, Mixed Models Analysis; LS Mean Difference = 0.4, 95% CI 2-sided [-0.5 to 1.4]
Statistical Analysis 3: Comparison: LY900014 vs LY900014 Postmeal; Total Daily Basal Insulin; Test type: Superiority; p = 0.693, Mixed Models Analysis; LS Mean Difference = -0.2, 95% CI 2-sided [-1.2 to 0.8]
Statistical Analysis 4: Comparison: Insulin Lispro (Humalog) vs LY900014; Total Daily Insulin Dose; Test type: Superiority; p = 0.625, Mixed Models Analysis; LS Mean Difference = 0.5, 95% CI 2-sided [-1.4 to 2.3]
Statistical Analysis 5: Comparison: Insulin Lispro (Humalog) vs LY900014 Postmeal; Total Daily Insulin Dose; Test type: Superiority; p = 0.758, Mixed Models Analysis; LS Mean Difference = -0.4, 95% CI 2-sided [-2.6 to 1.9]
Statistical Analysis 6: Comparison: LY900014 vs LY900014 Postmeal; Total Daily Insulin Dose; Test type: Superiority; p = 0.485, Mixed Models Analysis; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-3.1 to 1.5]

9. Secondary Outcome: Percentage of Participants With HbA1c < 7.0% and <7.5%
Description: Percentage of participants with HbA1c < 7.0% and <7.5% was analyzed using a longitudinal logistic regression with repeated measurements conducted by a generalized linear mixed model including independent variables of treatment, baseline HbA1c value, visit, baseline HbA1c-by-visit interaction, and treatment-by-visit interaction. An unstructured covariance structure was used.
Time Frame: Week 26
Population: All participants who were randomly assigned to study drug and had non-missing baseline value and at least one non-missing post-baseline value of the response variable.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Lispro (Humalog) | LY900014 | LY900014 Postmeal
Number analyzed (Participants) | 298 | 280 | 138
percentage of participants
  HbA1c <7% | 20.00 | 21.92 | 19.08
  HbA1c < 7.5% | 40.00 | 37.31 | 32.82
Statistical Analysis 1: Comparison: Insulin Lispro (Humalog) vs LY900014; HbA1c < 7%; Test type: Superiority; p = 0.396, Regression, Logistic; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.76 to 2.00]
Statistical Analysis 2: Comparison: Insulin Lispro (Humalog) vs LY900014 Postmeal; HbA1c < 7%; Test type: Superiority; p = 0.814, Regression, Logistic; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.49 to 1.75]
Statistical Analysis 3: Comparison: LY900014 vs LY900014 Postmeal; HbA1c < 7%; Test type: Superiority; p = 0.384, Regression, Logistic; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.39 to 1.43]
Statistical Analysis 4: Comparison: Insulin Lispro (Humalog) vs LY900014; HbA1c < 7.5%; Test type: Superiority; p = 0.400, Regression, Logistic; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.55 to 1.27]
Statistical Analysis 5: Comparison: Insulin Lispro (Humalog) vs LY900014 Postmeal; HbA1c < 7.5%; Test type: Superiority; p = 0.094, Regression, Logistic; Odds Ratio (OR) = 0.62, 95% CI 2-sided [0.36 to 1.08]
Statistical Analysis 6: Comparison: LY900014 vs LY900014 Postmeal; HbA1c < 7.5%; Test type: Superiority; p = 0.306, Regression, Logistic; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.43 to 1.31]

10. Secondary Outcome: Change From Baseline in 7-Point Self-Monitored Blood Glucose (SMBG) Values at Week 26
Description: Change from baseline in 7-point SMBG values were analyzed using MMRM and includes fixed class effects of treatment, strata (pooled country, type of basal insulin, and age group, and HbA1c stratum (≤8.0%, >8.0%)) baseline value, visit, and treatment-by-visit interaction. An unstructured covariance structure was used to model the within-participant errors.
Time Frame: Baseline, Week 26
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Insulin Lispro (Humalog) | LY900014 | LY900014 Postmeal
Number analyzed (Participants) | 298 | 280 | 138
mg/dL
  Morning Premeal - Fasting: number analyzed (Participants) | 265 | 247 | 122
  Morning Premeal - Fasting | 1.0 (2.78) | -3.4 (2.88) | -5.9 (4.11)
  Morning 1 hour Postmeal: number analyzed (Participants) | 263 | 239 | 117
  Morning 1 hour Postmeal | -3.2 (2.92) | -17.9 (3.06) | -9.8 (4.39)
  Midday Premeal: number analyzed (Participants) | 265 | 247 | 122
  Midday Premeal | -3.1 (3.06) | 2.5 (3.17) | -6.0 (4.52)
  Midday 1 hour Postmeal: number analyzed (Participants) | 262 | 237 | 120
  Midday 1 hour Postmeal | 0.9 (2.99) | -5.2 (3.14) | -1.5 (4.43)
  Evening Premeal: number analyzed (Participants) | 264 | 247 | 122
  Evening Premeal | 1.0 (3.18) | 4.6 (3.29) | 0.3 (4.69)
  Evening 1 hour Postmeal: number analyzed (Participants) | 261 | 234 | 118
  Evening 1 hour Postmeal | 6.9 (3.22) | -6.2 (3.39) | -3.9 (4.79)
  Bedtime: number analyzed (Participants) | 257 | 240 | 116
  Bedtime | -1.9 (3.03) | -2.3 (3.14) | -2.7 (4.53)

ADVERSE EVENTS:
Time Frame: From Lead-in to Safety Follow-up (up to 32 Weeks)
Description: All randomized participants who received at least one dose of study drug.
Groups:
- Humalog Lead-in: Participants received open-label insulin lispro (Humalog) administered subcutaneously (SC), using a unit for unit conversion or the dose was determined based on the investigator's clinical judgement.
- Humalog: Participants received 100 U/mL insulin lispro (Humalog) administered subcutaneously (SC), 0 to 2 minutes before each meal with once or twice daily basal insulin. Preprandial insulin doses were individualized and titrated according to protocol-defined targets.
Arm/Group | Humalog Lead-in | Humalog | LY900014 | LY900014 Postmeal
All-Cause Mortality (participants affected / at risk) | 0/751 | 0/298 | 0/280 | 0/138
Serious Adverse Events (participants affected / at risk) | 2/751 | 12/298 | 6/280 | 2/138
Other Adverse Events (participants affected / at risk) | 39/751 | 60/298 | 67/280 | 21/138
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Humalog Lead-in (N=751) | Humalog (N=298) | LY900014 (N=280) | LY900014 Postmeal (N=138)
Macroglossia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Complicated appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pilonidal cyst (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Reactive gastropathy (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemic coma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mental disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Humalog Lead-in (N=751) | Humalog (N=298) | LY900014 (N=280) | LY900014 Postmeal (N=138)
Vomiting (Gastrointestinal disorders) | 1 (1) | 9 (11) | 9 (10) | 3 (3)
Injection site reaction (General disorders) | 1 (1) | 0 (0) | 11 (14) | 2 (2)
Nasopharyngitis (Infections and infestations) | 21 (21) | 23 (30) | 28 (37) | 7 (9)
Rhinitis (Infections and infestations) | 7 (7) | 10 (10) | 6 (6) | 4 (5)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 16 (18) | 15 (17) | 2 (3)
Headache (Nervous system disorders) | 6 (6) | 13 (21) | 13 (22) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-04-30): https://cdn.clinicaltrials.gov/large-docs/19/NCT03740919/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-20): https://cdn.clinicaltrials.gov/large-docs/19/NCT03740919/SAP_001.pdf